CLINICAL TRIAL: NCT01129999
Title: The Comparative Efficacy of Cognitive-Behavioral Therapy (CBT) and Hypnotherapy (HT) for Smoking Cessation.
Brief Title: Cognitive-Behavioral Therapy and Hypnotherapy for Smoking Cessation
Acronym: CBT-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Anil Batra, Prof. Dr., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DKH-Studie VT-HT; 108368 (Other Grant/Funding Number: Deutsche Krebshilfe e.V.)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Smoking Cessation
Keywords: smoking cessation, CBT, hypnotherapy
MeSH Terms: conditions — Smoking Cessation; Color Vision Defects | interventions — Cognitive Behavioral Therapy; Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Hypnotherapy (Experimental)
  Interventions: Behavioral: Hypnotherapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — a cognitive-behavioral smoking cessation program; 6, weekly-held, group sessions (90 min each)
  Arms: Cognitive-Behavioral Therapy
Behavioral: Hypnotherapy — hypnotherapeutic smoking cessation program; 6, weekly-held, group sessions (90 min each)
  Other Names: hypnosis
  Arms: Hypnotherapy

SUMMARY:
Intensive cognitive-behaviour interventions (CBT) combined with pharmacotherapy for smoking cessation are well established and have been proved to be efficacious. Nevertheless, they yield only long-term abstinence rates about 35%. Considering the high interest of smokers in alternative medicine, the availability of a broad range of treatment methods, of which smokers choose an intervention according to their preferences, might contribute to improve treatment outcome. While hypnotherapy (HT) is an already widely promoted alternative method for aiding cessation, considerable methodological shortcomings of studies on this topic limit the interpretability of the results. In 2006, the German Academic Advisory Committee for Psychotherapy released new guidelines that included HT as an acceptable treatment for smoking cessation. The committee conceded, however, that conclusions concerning its efficacy are restricted due to the heterogeneity of findings. Hence, further well-designed studies are required to better test the efficacy of HT in comparison to accepted treatments. This randomised, controlled trial aims to compare the efficacy of CBT and HT for smoking cessation. Further, the influence of moderating variables will be investigated. It is hypothesized that 1) participants receiving CBT will evince higher abstinence rates than those receiving HT, 2) levels of nicotine dependence, self-efficacy and motivation to change will moderate the intervention effects and 3) participants with high levels of suggestibility will evince higher abstinence rates in the HT-intervention compared to participants with low levels of suggestibility. 220 adult healthy smokers will be randomized to receive either CBT or HT. Both programmes will be conducted in 6, weekly, 90-minute group sessions. Participants will be followed up at 1, 3, 6, 9 und 12 month post-treatment. Generalized estimating equation models will be conducted to analyse group differences on abstinence rates. The models will include the above mentioned moderator variables.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* smoking at least 10 cigarettes per day
* smoking at least for the past two years
* fluency in German language
* willing and able to give written informed consent

Exclusion Criteria:

* women: planned or current pregnancy or breast-feeding
* participation in a smoking cessation program within the last 6 months
* severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
12-months continuous smoking abstinence according to the Russell Standard (RS; West et al. 2005) | 12-months follow-up

SECONDARY OUTCOMES:
7-day point-prevalence smoking abstinence rates at 6- and 12-months follow-up | 12-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anil Batra, Prof., Study Director — University Hospital Tuebingen
Locations (1):
- University Hospital of Tuebingen Smoking Cessation Research Group, Tübingen, Germany

REFERENCES:
- [Derived] Batra A, Eck S, Riegel B, Friedrich S, Fuhr K, Torchalla I, Tonnies S. Hypnotherapy compared to cognitive-behavioral therapy for smoking cessation in a randomized controlled trial. Front Psychol. 2024 Feb 27;15:1330362. doi: 10.3389/fpsyg.2024.1330362. eCollection 2024. PMID 38476396